CLINICAL TRIAL: NCT04944849
Title: Reaction Time is Better in Digital Game Players
Brief Title: Reaction Time in Digital Game Players
Status: Completed | Type: Observational
Sponsor: Baskent University (Other)
Responsible Party: Principal Investigator, Nihan Ozunlu Pekyavas, Associated Proffesor, Baskent University
Other Study IDs: KA20/207
Record Dates: First submitted 2021-06-22; First posted 2021-06-30 (Actual); Last update posted 2022-01-14 (Actual); Status verified 2022-01

CONDITIONS: Computer Games
Keywords: digital game players; reaction time

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- digital gamer group: Individuals with computer use more than 14 hours a week were included in this group.
  Interventions: Diagnostic Test: Reaction Time Tests
- player group: Individuals with computer use less than 14 hours a week were included in this group.
  Interventions: Diagnostic Test: Reaction Time Tests

INTERVENTIONS:
Diagnostic Test: Reaction Time Tests — While doing our research, the reaction time test in the Human Benchmark application, where the reaction time to many different stimuli on the computer can be evaluated, the Aim Trainer test and the auditory reaction time tests at https://playback.fm/audio-reaction-time will be applied.

SUMMARY:
With the increasing use of computers in recent years, the effects of games have started to be discussed. Young people who play computers are exposed to many stimuli during the game and they react to these stimuli with reactions at various rates. In our study, we wanted to find out whether there is a significant difference in reaction time between young people who play computers more than 14 hours a week and those who do not.

DETAILED DESCRIPTION:
While doing our research, the reaction time test in the Human Benchmark application, where the reaction time to many different stimuli on the computer can be evaluated, the Aim Trainer test and the auditory reaction time tests at https://playback.fm/audio-reaction-time will be applied. The way the tests are applied; the first test will be separated as a trial and will not be included in the average. The next three tests will be averaged. Height, weight, smoking, use of antidepressants or stimulants, any ear or hearing problems, any eye disease, how many days a week and how much sports they do, the dominant side, whether they play digital and video games, for how long, what type of device (computer, tablet, phone), which games (League of legends, Player unknown's battlegrounds, World of Warcraft, Valorant, FIFA, PES, Call of duty, NBA, Counter strike:Global offensive CS:GO, other), how many hours a day and how many hours a week they play digital video games will be questioned whether they participate in the tournament with at least one of these games.

ELIGIBILITY:
Inclusion Criteria:

* male
* playing digital games for more than 2 years

Exclusion Criteria:

* female
* not having played any digital games for 2 years

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — male
Study Population: male individuals aged between 18-25 years who have been playing digital games for more than 2 years
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Visual reaction time | 15 minutes
  Visual reaction time will be evaluated with the Human Benchmark application. individuals will be asked to click on the specified area when the red light changes to green light. The test will be repeated 3 times and the average value will be recorded in ms.
Auditory reaction time | 15 minutes
  Auditory reaction time will be evaluated with the Aim Trainer test. individuals will be asked to click on the specified area when the red light changes to green light. The test will be repeated 3 times and the average value will be recorded in ms.

CONTACTS AND LOCATIONS:
Locations (1):
- Baskent University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided